CLINICAL TRIAL: NCT04475614
Title: Different Therapeutic Options for Burning Mouth Syndrome
Brief Title: Therapeutic Options for Treatment of Burning Mouth Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Assistant Professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01072018
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Burning Mouth Syndrome
Keywords: burning mouth syndrome; treatment
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Vitamin B Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- informative (No Intervention): The patients in this group received only verbal and written information about their condition.
- oral probiotics (Experimental): The patients in this group, beside verbal and written information about their condition, received also oral probiotics. They were instructed to melt one lozenge in the mouth in the evening, after tooth brushing and flossing, for one month.
  Interventions: Dietary Supplement: BioGaia Prodentis lozenges
- low level laser treatment (Experimental): The patients in this group, beside verbal and written information about their condition, received a total of ten low level laser treatments, for ten days consecutively excluding weekends.
  Interventions: Procedure: low level laser treatment with Ga-Al-As laser
- B-vitamin injections (Experimental): The patients in this group, beside verbal and written information about their condition, received a total of nine B vitamin injections, every other day, intra muscular.
  Interventions: Dietary Supplement: B vitamin injections (Neurobion, Merck, Darmstadt, Germany)

INTERVENTIONS:
Dietary Supplement: BioGaia Prodentis lozenges — oral probiotics
  Arms: oral probiotics
Procedure: low level laser treatment with Ga-Al-As laser — low level laser treatment
  Arms: low level laser treatment
Dietary Supplement: B vitamin injections (Neurobion, Merck, Darmstadt, Germany) — intra muscular vitamin injections
  Arms: B-vitamin injections

SUMMARY:
Burning mouth syndrome is a painful condition of unknown etiology that impairs the quality of life and does not have an adequate therapeutic option. The purpose of this study is to determine the most effective treatment option for burning mouth syndrome, among oral probiotics, low-level laser, B-vitamin injections and informative treatment only.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with burning mouth syndrome and excluded local and systemic causes

Exclusion Criteria:

* patients who have received treatment for burning mouth earlier
* patients with local or systemic causes of burning mouth

Ages: 39 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in the patient's quality of life using Oral Health Impact Profile 14 questionnaire (OHIP-14) | up to two months (follow up was one month after the end of treatment, in each patient)
  change in the patient's quality of life determined by self-perceived quality of life questionnaire (Oral Health Impact Profile; OHIP-14)

SECONDARY OUTCOMES:
Change in subjective burning symptoms | up to two months (follow up was one month after the end of treatment, in each patient)
  change of patient's subjective burning symptoms measured on visual analogue scale (VAS) grading from 0 to 10 (0- without burning, 10- the worst possible burning)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No